CLINICAL TRIAL: NCT02738008
Title: A Multicenter, Extension Study of the Safety and Efficacy of Multi-dose Intravenous ARC-520 in Combination With Entecavir or Tenofovir in Patients With Chronic Hepatitis B Virus (HBV) Infection
Brief Title: Extension Study of the Safety and Efficacy of Multi-dose Intravenous ARC-520 in Patients With Chronic Hepatitis B (HBV) Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision to discontinue trial
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Heparc-2007; 2014-004201-33 (EudraCT Number)
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — ARC-520; entecavir; Tenofovir; Histamine Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ARC-520 Injection (Experimental): Multiple administrations of ARC-520 starting at a dose level of 2 mg/kg, plus entecavir (0.5 or 1.0 mg/day) or tenofovir (300 mg/day)
  Interventions: Drug: ARC-520 Injection; Drug: entecavir; Drug: tenofovir; Drug: antihistamine

INTERVENTIONS:
Drug: ARC-520 Injection — IV injection
Drug: entecavir — All participants will take entecavir or tenofovir throughout the study. Participants will be instructed to take their medication daily.
Drug: tenofovir — All participants will take entecavir or tenofovir throughout the study. Participants will be instructed to take their medication daily.
Drug: antihistamine — All participants will be pretreated with an oral antihistamine. The antihistamine used should in general be an H1>H2 receptor blocker and would include diphenhydramine 50 mg, cetirizine 10 mg, chlorpheniramine 8 mg or hydroxyzine 50 mg. The Investigator is free to choose any of these antihistamines available locally and consistent with their country's Marketing Authorisation.

SUMMARY:
Chronic HBV patients will receive 9 doses of open-label ARC-520 once every 4 weeks and be evaluated for safety and efficacy.

DETAILED DESCRIPTION:
Open-label, multi-center extension study of intravenous ARC-520 in combination with entecavir or tenofovir in patients with chronic HBV infection. Patients who successfully completed the Heparc-2002 (NCT02604199) and Heparc-2003 (NCT02604212) studies and responded to therapy are eligible to participate. Responders are defined as patients who showed a ½ log or greater reduction in their serum Hepatitis B Surface Antigen (HBsAg) levels from baseline to day 71 ± 3 days of the primary Heparc-2002 and Heparc-2003 studies. Patients who have signed a Human Research Ethics Committee approved informed consent and have met all of the protocol eligibility criteria will continue receiving daily oral entecavir or tenofovir and intravenous (IV) injections of ARC-520. Study visits will occur once every 4 weeks for a total of 9 visits for monitoring and ARC-520 administration.

Patients will undergo the following evaluations at regular intervals during the study: medical history, physical examinations, vital sign measurements (blood pressure, heart rate, respiratory rate and temperature), weight, adverse events (AEs), 12-lead electrocardiograms (ECGs), concomitant medications, blood sample collection for hematology, coagulation, chemistry, creatine kinase, troponin, hemoglobin A1c, exploratory pharmacodynamic (PD) measures, urinalysis, HBV serology, immunogenicity, and pregnancy testing for females of childbearing potential. Patients will be monitored for HBV virology, AEs, and exploratory PD measures for a total of 24 weeks after the last dose of ARC-520.

ELIGIBILITY:
Inclusion Criteria:

* Patient showed a ½ log or greater reduction in serum HBsAg levels from baseline to Day 71 ± 3 days or Day 99 ± 3 days in the primary Heparc-2002 or Heparc-2003 study.
* Able to have first dose within 2 months of day 113 end-of-study visit in the primary Heparc-2002 or Heparc-2003 study.
* Able to provide written informed consent prior to the performance of any study specific procedures.
* Have no abnormalities in 12-lead ECG assessment that, in the opinion of the investigator, may compromise patient safety
* Willing and able to comply with all study assessments and adhere to the protocol schedule.
* Have no new abnormal finding of clinical relevance at the screening evaluation.
* Using 2 effective methods of contraception (double barrier contraception or hormonal contraceptive along with a barrier contraceptive) (both male and female partners) during the study and for 3 months following the last dose of (ARC 520).

Exclusion Criteria:

* Pregnant or lactating.
* Acute signs of hepatitis/other infection within 4 weeks of screening and/or at the screening examination.
* Use of prescription medication (including anticoagulants) within 14 days prior to administration of ARC-520.
* Has had major surgery within 3 months of screening.
* Has evidence of severe systemic acute inflammation, sepsis, or hemolysis.
* Diagnosed with a significant psychiatric disorder that would prevent participation in the study.
* Unable or unwilling to return for all scheduled study visits.
* Has any other condition that, in the opinion of the investigator, would render the patient unsuitable for enrollment, or could interfere with his/her participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Research Site 1, Hong Kong, China
- Research Site 2, Leipzig, Germany
- South Korea (4):
  - Research Site 3, Busan
  - Research Site 5, Incheon
  - Research Site 4, Seoul
  - Research Site 6, Seoul

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in participants who successfully completed the primary studies Heparc-2002 (NCT02604199) and Heparc-2003 (NCT02604212) through Day 113 and responded to therapy, except for those who achieved loss of Hepatitis B Surface Antigen (HBsAg) during the primary study.
Pre-assignment Details: No participants were enrolled from the Heparc-2002 or Heparc-2003 placebo groups.
Groups:
- Heparc-2002: ARC-520 1.0 mg/kg: ARC-520 2.0 mg/kg administered by intravenous (IV) infusion to participants previously enrolled in the Heparc-2002 study and receiving ARC-520 1.0 mg/kg. Participants continued their ongoing entecavir therapy (0.5 or 1.0 mg/day) or tenofovir therapy (300 mg/day).
- Heparc-2002: ARC-520 2.0 mg/kg: ARC-520 2.0 mg/kg administered by IV infusion to participants previously enrolled in the Heparc-2002 study and receiving ARC-520 2.0 mg/kg. Participants continued their ongoing entecavir therapy (0.5 or 1.0 mg/day) or tenofovir therapy (300 mg/day).
- Heparc-2003: ARC-520 2.0 mg/kg: ARC-520 2.0 mg/kg administered by IV infusion to participants previously enrolled in the Heparc-2003 study and receiving ARC-520 2.0 mg/kg. Participants continued their ongoing entecavir therapy (0.5 or 1.0 mg/day) or tenofovir therapy (300 mg/day).
Period: Overall Study
Arm/Group | Heparc-2002: ARC-520 1.0 mg/kg | Heparc-2002: ARC-520 2.0 mg/kg | Heparc-2003: ARC-520 2.0 mg/kg
Started | 1 | 6 | 5
Completed | 0 | 0 | 0
Not Completed | 1 | 6 | 5
Not completed — Study Terminated by Sponsor | 1 | 5 | 3
Not completed — Adverse Event | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Heparc-2002: ARC-520 1.0 mg/kg: ARC-520 2.0 mg/kg administered by IV infusion to participants previously enrolled in the Heparc-2002 study and receiving ARC-520 1.0 mg/kg. Participants continued their ongoing entecavir therapy (0.5 or 1.0 mg/day) or tenofovir therapy (300 mg/day).
- Total: Total of all reporting groups
Arm/Group | Heparc-2002: ARC-520 1.0 mg/kg | Heparc-2002: ARC-520 2.0 mg/kg | Heparc-2003: ARC-520 2.0 mg/kg | Total
Number analyzed (Participants) | 1 | 6 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 5 | 5 | 11
  >=65 years | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 2 | 7
  Male | 1 | 1 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Initial Responders to ARC-520 Therapy Achieving a 1-log Reduction in HBsAg at Week 36 Compared to Baseline
Description: Initial responders are defined as participants who showed a ½ log or greater reduction in their serum HBsAg levels from baseline to Day 71 ± 3 days of the primary Heparc-2002 and Heparc-2003 studies, where baseline is defined as the average of pre-dose values.
Time Frame: Baseline, Week 36
Population: The study was terminated prior to any participant reaching Week 36 of treatment; therefore, this outcome measure could not be analyzed.
Arm/Group | Heparc-2002: ARC-520 1.0 mg/kg | Heparc-2002: ARC-520 2.0 mg/kg | Heparc-2003: ARC-520 2.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence which does not necessarily have a causal relationship with this treatment. An SAE is any AE that: results in death; is life-threatening; requires inpatient hospitalization or prolongation of an existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or is a medically important event or reaction. A TEAE was defined as an AE that was not present prior to the first study medication administration and started at/after the time of initiation of administration of study medication, or an AE which was present prior to initiation of study medication administration, which increased in severity after study medication administration.
Time Frame: From first dose of study drug up to 28 weeks of treatment, plus up to 24 weeks of follow-up
Population: Safety Population: all participants who received at least 1 dose of study medication and had at least 1 post-dose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Heparc-2002: ARC-520 1.0 mg/kg | Heparc-2002: ARC-520 2.0 mg/kg | Heparc-2003: ARC-520 2.0 mg/kg
Number analyzed (Participants) | 1 | 6 | 5
Participants
  AEs | 1 | 4 | 4
  SAEs | 0 | 0 | 0

3. Secondary Outcome: Percentage of Initial Responders to ARC-520 Therapy With HBsAg Loss (Qualitative) Compared to Baseline Over Time
Description: The qualitative HBsAg assay gives a binary result, positive or negative. Baseline is defined as the average of the pre-dose values in the primary Heparc-2002 and Heparc-2003 studies.
Time Frame: Baseline, Weeks 36, 48, and 60
Population: as for outcome 1
Arm/Group | Heparc-2002: ARC-520 1.0 mg/kg | Heparc-2002: ARC-520 2.0 mg/kg | Heparc-2003: ARC-520 2.0 mg/kg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 28 weeks of treatment, plus up to 24 weeks of follow-up
Description: TEAEs are presented. A TEAE was defined as an AE that was not present prior to the first study medication administration and started at/after the time of initiation of administration of study medication, or an AE which was present prior to initiation of study medication administration, which increased in severity after study medication administration.
Arm/Group | Heparc-2002: ARC-520 1.0 mg/kg | Heparc-2002: ARC-520 2.0 mg/kg | Heparc-2003: ARC-520 2.0 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 1/1 | 4/6 | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Heparc-2002: ARC-520 1.0 mg/kg (N=1) | Heparc-2002: ARC-520 2.0 mg/kg (N=6) | Heparc-2003: ARC-520 2.0 mg/kg (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Chest discomfort (General disorders) | 0 | 0 | 2
Chills (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hyposaesthesia (Nervous system disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
The decision to discontinue development of ARC-EXl-containing programs was not due to any safety findings in clinical studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No